CLINICAL TRIAL: NCT06918314
Title: The Effect of Blood Flow Restriction Exercise on Muscle Oxygenation and Lactate Levels in Elite Athletes: A Comparative Study
Brief Title: "How Blood Flow Restriction Exercise Affects Muscle Oxygenation and Lactate in Elite Athletes"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator PhD Physiotherapist Burcin Ugur Tosun, Eastern Mediterranean University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-177
Record Dates: First submitted 2025-03-12; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Blood Flow Restriction Training; Muscle Oxygenation; Physiological Adaptations
Keywords: elite athletes; moxy; bfr; aerobic exercise; treadmill; Blood Lactate Levels

STUDY DESIGN:
Intervention Model Description: "This study aims to compare two distinct groups: healthy sedentary male individuals and healthy elite male athletes. The research will focus on various physiological and performance-related parameters to examine the differences between these groups in terms of muscle function, cardiovascular efficiency, metabolic responses, and overall physical fitness. By analyzing these factors, the study seeks to provide valuable insights into the impact of regular high-intensity training on physical health and performance, as well as how a sedentary lifestyle affects these parameters. The findings may contribute to a better understanding of training adaptations and the physiological characteristics distinguishing elite athletes from their sedentary counterparts."
Who Masked: Participant
Masking Description: Healthy Sedentary Male Individuals: These participants are physically inactive or engage in minimal physical activity. They do not follow a structured exercise regimen and have no history of professional or competitive sports participation. They are in good general health, with no chronic diseases or musculoskeletal disorders that could affect the study outcomes.
  Healthy Elite Male Athletes: These participants are actively involved in elite-level athletics, following a structured and high-intensity training program. They have extensive experience in competitive sports, particularly in track and field disciplines. They are in optimal physical condition, with well-developed cardiovascular and musculoskeletal systems, and no history of major injuries or health conditions that could impact their performance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Elite Male Athletes (Experimental): These participants are physically inactive or engage in minimal physical activity. They do not follow a structured exercise regimen and have no history of professional or competitive sports participation. They are in good general health, with no chronic diseases or musculoskeletal disorders that could affect the study outcomes.
  Interventions: Device: Blood Flow Restriction Kaatsu Training Device
- Healthy Sedentary Male Individuals (Active Comparator): These participants are actively involved in elite-level athletics, following a structured and high-intensity training program. They have extensive experience in competitive sports, particularly in track and field disciplines. They are in optimal physical condition, with well-developed cardiovascular and musculoskeletal systems, and no history of major injuries or health conditions that could impact their performance.
  Interventions: Device: Blood Flow Restriction Kaatsu Training Device

INTERVENTIONS:
Device: Blood Flow Restriction Kaatsu Training Device — The Blood Flow Restriction (BFR) intervention uses a pneumatic cuff to partially restrict arterial and fully restrict venous blood flow, creating a hypoxic environment that enhances muscle activation and strength at low exercise intensities. In this study, BFR will be applied intermittently during low-intensity treadmill walking with controlled pressure adjustments.
  The Moxy Muscle Oxygen Monitor is a non-invasive NIRS device that measures muscle oxygen saturation (SmO₂) and total hemoglobin (THb). Placed on the quadriceps femoris muscle, it will track oxygenation changes before, during, and after BFR exercise, helping assess muscle metabolism and performance adaptations.
  Other Names: Moxy Muscle Oxygenation

SUMMARY:
This study investigates the effects of blood flow restriction (BFR) training combined with low-intensity aerobic exercise on muscle oxygenation, total hemoglobin (THb), and blood lactate levels in elite athletes, comparing them with healthy sedentary individuals. BFR training, which partially restricts arterial and fully restricts venous blood flow using a pneumatic cuff, creates a hypoxic environment, leading to muscle strength and endurance improvements with lower-intensity exercise. The study aims to determine whether BFR-induced occlusion enhances muscle adaptation and how these physiological responses differ between elite athletes and sedentary individuals.

DETAILED DESCRIPTION:
This comparative cross-sectional study aims to examine the acute physiological responses to low-intensity aerobic exercise combined with blood flow restriction (BFR) training in elite male track and field athletes versus sedentary individuals. The primary focus is on changes in muscle oxygenation, total hemoglobin (THb), and blood lactate concentrations.

BFR is applied via a pneumatic cuff that partially restricts arterial and fully restricts venous return, thereby creating a localized hypoxic environment. This method has been shown to induce strength and endurance adaptations comparable to high-intensity training, even when performed at low intensities.

Near-infrared spectroscopy (NIRS) via the Moxy Muscle Oxygen Monitor will be used to assess muscle oxygenation parameters in real-time. Blood lactate levels will be measured through capillary sampling before and after exercise. Additional physiological parameters including heart rate, blood pressure, and respiratory rate will also be monitored.

The study compares two groups with distinct physical activity backgrounds, intending to elucidate potential differences in physiological adaptation to BFR. All measurements will be carried out in a controlled lab environment using validated instruments. Statistical analyses will be performed using SPSS software, with appropriate parametric or non-parametric methods depending on data distribution.

The results may contribute to a deeper understanding of BFR training mechanisms and guide tailored conditioning strategies for both athletic and sedentary populations.

ELIGIBILITY:
Eligibility Criteria:

Participants will be included or excluded based on the following conditions:

Inclusion Criteria:

Willingness to participate in the study

Male individuals aged 15-18 years

Sedentary status for control group participants (<600 MET-min/week according to the International Physical Activity Questionnaire - Short Form)

Body mass index (BMI) <25 kg/m²

Licensed track and field athlete for the study group

At least 3 years of experience as a licensed sprint athlete

No history of sports injury in the last 6 months

Exclusion Criteria:

Presence of open wounds or infection in the lower extremities

Leg pain, varicose veins, or thrombophlebitis

Diabetes or a history of cardiovascular disease

Smoking and/or alcohol consumption

Presence of respiratory distress

Bilateral lower extremity pain and edema

Incompatibility with the blood flow restriction (BFR) device

Presence of diseases causing endothelial dysfunction (e.g., hypertension, cardiovascular diseases, neurological disorders, systemic inflammation, obesity, diabetes, atherosclerosis)

History of deep vein thrombosis (DVT) or peripheral vascular disease

Presence of acute infection

History of cancer

Surgical operation due to trauma within the last 6 months

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Change in muscle oxygenation (SmO₂) measured by Moxy Muscle Oxygen Monitor (Near-Infrared Spectroscopy - NIRS) | Over a period of 2 months
  Muscle oxygenation (SmO₂) will be assessed using the Moxy Muscle Oxygen Monitor, a validated NIRS-based device placed on the vastus lateralis muscle. Measurements will be taken pre- and post-exercise across multiple sessions to observe acute and cumulative responses.Unit of Measure: Percentage (%)
Change in blood lactate concentration measured by portable lactate analyzer (e.g., Lactate Scout+) | Immediately before and 3 minutes after each exercise session over a 2-month period
  Capillary blood samples will be collected from the fingertip immediately before and 3 minutes after low-intensity aerobic exercise. Lactate levels will be analyzed using a validated point-of-care lactate analyzer to assess the metabolic response to BFR training.Unit of Measure: mmol/L
Change in body fat percentage measured by Bioelectrical Impedance Analysis (TANITA BIA device) | Over a period of 2 months
  Body fat percentage will be assessed using a validated TANITA BIA device to evaluate changes in body composition.
Change in muscle mass measured by Bioelectrical Impedance Analysis (TANITA BIA device) | Baseline and end of 2-month intervention
  Muscle mass will be assessed using a TANITA BIA device to track training-induced adaptations. Unit of Measure: Kilograms (kg)
Change in Body Mass Index (BMI) measured by Bioelectrical Impedance Analysis (TANITA BIA device) | Baseline and end of 2-month intervention
  BMI will be calculated from height and weight data provided by the TANITA BIA device to observe general body composition trends. Unit of Measure: kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: gulhan yılmaz gokmen, Assoc. Prof., Study Director — "Bandırma Onyedi Eylül University, Faculty of Health Sciences"
Locations (1):
- Burcin Ugur Tosun, Famagusta, Cyprus